CLINICAL TRIAL: NCT03561285
Title: Antiphospholipid Antibodies & Osteopontin as Risk Factors for Cerebrovascular Stroke in Young Adults
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sally Samir Youssef, Investigator, Assiut University
Other Study IDs: 17200187
Record Dates: First submitted 2018-04-13; First posted 2018-06-19 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Stroke in Young Adults

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke with antiphospholipid
  Interventions: Diagnostic Test: antiphospholipid Abs
- stroke without antiphospholipid
  Interventions: Diagnostic Test: antiphospholipid Abs

INTERVENTIONS:
Diagnostic Test: antiphospholipid Abs — Laboratory test

SUMMARY:
The burden of stroke is increasing in many low- and middle income countries.(1) Around 10% of all thrombotic cerebrovascular events (CVE) occur in young population defined as younger than 50 years old (2)

In the majority of these patients, the cause of the ischaemic stroke remains undetermined.(3) Arterial thrombosis is a major clinical manifestation of the antiphospholipid syndrome (APS), an autoimmune condition characterised by thrombotic events and/or pregnancy morbidity with persistently positive antiphospholipid antibodies (aPL) (4).

Considering all patients with cerebral ischaemia, the prevalence of aPL seems rather high in young adults, who might constitute a subgroup at high risk for recurrence.(5)

Through the support of the Antiphospholipid Syndrome Alliance for Clinical Trials and International Networking (APS ACTION), a systematic review aiming to estimate the frequency of clinically significant aPL profiles in the general population (no age limit) was completed. (6)

The pathogenesis of ischemic stroke is complex, and several studies documented hypercoagulable states as a significant mechanism underlying stroke. (8).

The latter include protein C, protein S, or antithrombin III deficiencies, activated protein C resistance and anti-phospholipid antibodies (aPLA), including anticardiolipin (aCL) antibodies or lupus anticoagulant (LAC), which influence stroke susceptibility owing to their capacity to disturb normal hemostatic mechanisms (9).

While aPLA are clinically associated with a state of hypercoagulation and prothrombotic disorders, the exact mechanism underlying their prothrombotic effects remains unknown (10).

aPLA are detected either functionally, owing to their ability to prolong coagulation time in a phospholipid-dependent coagulation test (LAC), or by measuring specific [anticardiolipin (aCL) and antiphosphatidylserine (aPS)] antibodies by specific immunoassays, using anionic phospholipids as antigens (11).

The contribution of LAC to the overall risk of both venous and arterial thrombosis, including ischemic stroke, is now well recognized (12).

While the contribution of aPLA (including LAC and aCL antibodies) to thrombosis is well established, their role as independent risk factors in the pathogenesis of ischemic stroke yielded apparently conflicting results. (13).

These conflicting results could be explained by differences in ethnic origin , inherent variation in aPLA levels and in the failure in some studies to account for the contribution of covariates (14).

Osteopontin (OPN) was first identified as a protein involved in bone remodelling, but later also shown to have important immunological roles. (15).

ELIGIBILITY:
Inclusion Criteria:

* A study was included if it reported on the laboratory investigation of any aPL and confirmed CVE
* Included patients aged <50 years

Exclusion Criteria:

* Exclusion criteria included non-atherosclerotic causes, rheumatic heart disease, ventricular arrhythmias, uncompensated heart failure, stroke secondary to atrial fibrillation, hematoma, brain tumors, accidental or iatrogenic stroke, arterial malformation and recent acute myocardial infarction. Information on cardiovascular and cerebrovascular risk factors will be obtained at baseline.
* Cardiovascular disease will positive if subjects reported a history of heart disease or stroke, whereas diabetes will be assessed according to fasting blood glucose and/or use of glucose-lowering drugs (including insulin).

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: stroke patients less than 50 years old
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Stroke patients with APs | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eman Abbas El kady, Prof., Study Director — Investigator
Locations (1):
- Assiut University Hospital, Asyut, Egypt